CLINICAL TRIAL: NCT02448953
Title: Comparison of Lymph Node Dissection Results and Prognosis in Thoracic Esophageal Carcinoma Without Cervical Lymph Node Involvement: Two-field Versus Three-field Lymph Node Dissection
Brief Title: Two-field Versus Three-field Lymphadenectomy in Thoracic Esophageal Carcinoma Without Cervical Lymph Node Involvement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Henan Cancer Hospital (Other Government); Hebei Medical University Fourth Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other); Fujian Cancer Hospital (Other Government); Liaoning Cancer Hospital & Institute (Other); Zhejiang Cancer Hospital (Other); Tongji Hospital (Other); Tang-Du Hospital (Other); Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jie He, president, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NKTRDP-2015BAI12B08-03
Record Dates: First submitted 2015-05-08; First posted 2015-05-20 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Esophageal Cancer
Keywords: Without cervical lymph node involvement
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- negative lymph node (Active Comparator): lymph node along the right recurrent laryngeal nerve should be confirmed negative by intraoperative frozen pathology examination
  Interventions: Procedure: Two-field lymphadenectomy; Procedure: Three-field lymphadenectomy
- positive lymph node (Active Comparator): lymph node along the right recurrent laryngeal nerve should be confirmed negative by intraoperative frozen pathology examination
  Interventions: Procedure: Three-field lymphadenectomy

INTERVENTIONS:
Procedure: Two-field lymphadenectomy — Thoracic-upper abdominal two-field lymphadenectomy
  Arms: negative lymph node
Procedure: Three-field lymphadenectomy — Cervical-thoracic-upper abdominal three-field completely lymphadenectomy

SUMMARY:
The purpose of this study is to compare the lymph node dissection results and prognosis in thoracic esophageal carcinoma patients without cervical lymph node involvement by preoperative CT and/or ultrasound treated by two-field lymphadenectomy or three-field lymphadenectomy.Another purpose of this study is to clarify whether the lymph node along the right recurrent laryngeal nerve can be taken as the sentinel lymph node which is able to indicate neck lymph node metastasis and necessity for three-field lymphadenectomy.

DETAILED DESCRIPTION:
Esophageal carcinoma is a prevalent and aggressive malignant disease with poor prognosis in China. Complete surgical resection with systemic lymph node dissection remains the most effective treatment method for this malignancy. Although tree-field lymph node dissection was reported to be effective in improving long-term survival in Japan,there is no enough evidences yet to demonstrate that three field lymph node dissection is superior to two field lymph node dissection in reducing postoperative recurrence and improving long-term survival. In this study, the dissection of lymph node adjacent to the right recurrent laryngeal nerve would be performed and examined routinely by intraoperative frozen-section. If the lymph node is positive, three field lymph node dissection(Cervical-thoracic-upper abdominal lymphadenectomy) will be performed, if negative, the patients will be randomly assigned either to three-field lymphadenectomy group or two-field lymphadenectomy group. The purpose of this large scale multi-center trial is to compare the lymph node dissection results and prognosis in thoracic esophageal carcinoma without cervical lymph node involvement treated by three-field lymphadenectomy or two-field lymphadenectomy and clarify whether the lymph node along the right recurrent laryngeal nerve could be taken as sentinel lymph node indicating neck lymph node metastasis and necessity of three-field lymphadenectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed squamous cell esophageal cancer, without any previous anti-tumor therapy;
2. Preoperative clinical TNM stage：cT1b-3N0-1M0;
3. Adequate cardiopulmonary, liver, brain and kidney functions for esophagectomy either via right thoracotomy or VATS;
4. No evidence of suspicious neck lymph node metastasis (LN short diameter < 0.8cm or LN short/long diameter <0.65 by cervical CT and/or ultrasound);
5. Willing to participate the clinical trial and sign the informed consent before being enrolled into clinical trail

Exclusion Criteria:

1. Previous use of anti-cancer therapy;
2. Preoperative clinical TNM stage: N2-3 or M1;
3. Inadequate cardiopulmonary,liver, brain and kidney function for surgery;
4. Previous malignancy history.
5. Suspicious neck lymph node metastasis (LN short diameter ≧0.8cm or LN short/long diameter ≧0.65 by cervical CT and/or ultrasound);
6. Unwilling to participate the clinical trial and refuse to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 786 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Long term survival | 5 years

SECONDARY OUTCOMES:
Disease free survival | 5 years
Locoregional recurrence | 5 years
Postoperative complications | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jie He, MD,PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Mao Y, Liu S, Han Y, Guo S, Chen C, Gao S, Hao A, Duan H, Fang W, Zhang R, Yu Z, Fu X, Li X, Wang Q, Tan L, Li Z, Li Y, Zhang Z, Wei W, Fang Y, Fu D, Wei X, Yuan L, Muhammad S, He J. Three-field vs two-field lymphadenectomy in thoracic ESCC patients: a multicenter randomized study (NST 1503). J Natl Cancer Cent. 2025 Jan 14;5(2):203-211. doi: 10.1016/j.jncc.2025.01.002. eCollection 2025 Apr. PMID 40265094